CLINICAL TRIAL: NCT00245427
Title: Outcomes of Patients Not Responding to Outpatient Macrolide or b-Lactam Therapy for the Treatment of Community Acquired Pneumonia: Expansion to Include Acute Exacerbations of Chronic Bronchitis and Acute Sinusitis
Brief Title: Outcomes of Patients Not Responding to Antibiotics in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CPL Associates (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: HMR3647A-6012
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Sinusitis; Bronchitis, Chronic; Pneumonia, Bacterial
Keywords: beta-lactam; macrolide; antibiotics
MeSH Terms: conditions — Sinusitis; Bronchitis, Chronic; Pneumonia, Bacterial

ARMS (2):
- 1 All macrolide antibiotics (Other)
  Interventions: Drug: all macrolide antibiotics
- 2 All beta lactam antibiotics (Other)
  Interventions: Drug: all beta-lactam antibiotics

INTERVENTIONS:
Drug: all macrolide antibiotics — Varies based on antibiotic
  Arms: 1 All macrolide antibiotics
Drug: all beta-lactam antibiotics — Varies based on antibiotic
  Arms: 2 All beta lactam antibiotics

SUMMARY:
A study to report the outcomes of patients who fail to respond to beta-lactam and macrolide antibiotics in the community

DETAILED DESCRIPTION:
To document and describe the clinical, microbiological, and pharmacoeconomic outcomes of two hundred patients who failed to respond to outpatient macrolide or beta-lactam therapy. Evaluable patients must have a positive culture obtained after they failed their initial macrolide or beta-lactam. The isolated pathogen must have a known MIC to the antibiotic class they failed to respond to (i.e. macrolide or b-lactam). The isolate must be available to be sent to the central laboratory for MIC testing

ELIGIBILITY:
Inclusion Criteria:

Patients who have failed to respond to at least three (ABECB and CAP) or five (AMS/ABRS/AECRS) days of macrolide or b-lactam therapy meeting all of the protocol criteria for acute bacterial exacerbations on chronic bronchitis(ABECB), community acquired pneumonia(CAP) and acute maxillary sinusitis(AMS) will be eligible for enrollment. All patients, whether enrolled retrospectively or concurrently, must have a positive culture. The pathogenic bacteria must be identified by a local laboratory and have a known susceptibility to the antibiotic class the patient failed to respond to (i.e. macrolide or b-lactam). The isolate must be sent to the Study Coordinating Center for precise MIC determination.

Exclusion Criteria:

Patients presenting with any of the following will not be included in the study:

1. Life expectancy <3 months from underlying disease
2. Underlying lung carcinoma
3. Cystic fibrosis

Max Age: 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-12; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Clinical outcome | varies

SECONDARY OUTCOMES:
PK/PD pharmacoeconomics | varies

CONTACTS AND LOCATIONS:
Overall Officials: Jerome J Schentag, Pharm.D., Principal Investigator — State University of NY at Buffalo; Joseph Paladino, Pharm.D., Study Director — State University of NY at Buffalo
Locations (1):
- Deaconess Medical School, Spokane, Washington, United States

REFERENCES:
- See also: Related Info — http://www.cplassociates.com